CLINICAL TRIAL: NCT05515900
Title: The Roles of HMB and Sodium in Blood Pressure Regulation and Gut Microbiome
Brief Title: Salt and HMB Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1810996
Record Dates: First submitted 2022-07-20; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Blood Pressure
MeSH Terms: interventions — Sodium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sodium active, HMB active (Experimental): The subjects in this group will take sodium pills of 2,000 mg/day from baseline to week 8, and take HMB pills of 3 g/day from week 5 to week 8 while on reduced-sodium diet.
  Interventions: Dietary Supplement: Sodium; Dietary Supplement: HMB
- Sodium active, HMB placebo (Experimental): The subjects in this group will take sodium pills of 2,000 mg/day from baseline to week 8, and take placebo pills of 3 g/day from week 5 to week 8 while on reduced-sodium diet.
  Interventions: Dietary Supplement: Sodium
- Sodium placebo, HMB active (Experimental): The subjects in this group will take placebo pills from baseline to week 8, and take HMB pills of 3 g/day from week 5 to week 8 while on reduced-sodium diet.
  Interventions: Dietary Supplement: HMB
- Sodium placebo, HMB placebo (Placebo Comparator): The subjects in this group will take placebo pills from baseline to week 8 while on reduced-sodium diet.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Sodium — Daily sodium supplementation of 2000 mg.
  Arms: Sodium active, HMB active; Sodium active, HMB placebo
Dietary Supplement: HMB — Daily HMB supplementation of 3 g.
  Arms: Sodium active, HMB active; Sodium placebo, HMB active
Other: Placebo — Placebo pills that will be identical to sodium or HMB supplementations
  Arms: Sodium placebo, HMB placebo

SUMMARY:
Hypertension affects one-third of adults in the US. High salt diet is a key risk factor for elevated blood pressure (BP). The associations of gut microbiome with high salt diet and hypertension have been established in both animal and human studies. However, the underlying biological mechanisms linking sodium to BP elevation and gut microbiome alteration are not clear. Increasing evidence supports a pivotal role of leucine metabolism in hypertension. Leucine is initially catalyzed by the branched-chain amino acid aminotransferase enzyme (BCAT), producing α-ketoisocaproate (α-KIC), which can be further metabolized to β-hydroxy-β-methylbutyrate (HMB). Leucine/α-KIC/HMB metabolism pathway shows a promising involvement in the relationships among salt, gut microbiome, and elevated BP. Preliminary studies show that dietary sodium reduction increases circulating HMB, which is further associated with reduced BP, and that HMB treatment decreases Firmicutes/Bacteroidetes ratio, and increases α-diversity and gut microbiota-derived short-chain fatty acids (SCFAs). However, the leucine/α-KIC/HMB metabolism pathway has never been targeted in human studies. To establish causality, I propose a double-blind, two-stage randomized, placebo-controlled trial of sodium and HMB supplements for the following specific aims: Aim 1 will determine the effect of sodium supplement on leucine/α-KIC/HMB metabolism pathway. Aim 2 will determine the effect of HMB supplement on office BP and 24-hour ambulatory BP (Aim 2a), and α- and β-diversities and Firmicutes/Bacteroidetes ratio (Aim 2b). Secondary Aim will test the hypothesis that HMB supplement could partially block the detrimental effects of sodium intake on BP and gut microbiota. The proposed project would help to uncover the role of leucine/α-KIC/HMB metabolism pathway in salt-induced hypertension and the alteration in gut microbiome. Most importantly, the project will provide the training opportunities for me as a junior faculty, to study the new area of gut microbiome, acquire new experience and skills to conduct human trials. In addition, this project will generate rich preliminary data on the role of leucine/α-KIC/HMB metabolism pathway in salt-induced BP elevation, and test the feasibility for developing future NIH R01 project.

ELIGIBILITY:
Inclusion Criteria:

* normotensive [SBP<140 mmHg and diastolic BP (DBP)<90 mmHg];
* self-identified black or white; c. aged from 18 to 65 years.

Exclusion Criteria:

* taking medication that would affect BP or gut microbiome;
* being pregnant;
* with health conditions that would compromise sodium handling.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Leucine/α-KIC/HMB metabolism | 4 weeks
  Changes in blood levels of metabolites leucine, α-KIC, and HMB from baseline to week 4.
Blood pressure | 4 weeks
  Changes in systolic and diastolic blood pressure from week 5 to week 8.
Gut microbiome | 4 weeks
  Changes in the composition of gut microbiome from week 5 to week 8.

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided